CLINICAL TRIAL: NCT04081311
Title: A Comparison of the Efficacy of Interdental Floss to Water Flosser Around Dental Implants in Maintenance Patients: a Randomized Controlled Trial
Brief Title: A Comparison of the Efficacy of Interdental Floss to Water Flosser Around Dental Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H2019:298
Record Dates: First submitted 2019-09-04; First posted 2019-09-09 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Implant Site Bleeding
Keywords: dental implants; water flosser

STUDY DESIGN:
Intervention Model Description: Randomized, controlled clinical trial in a single center.
Who Masked: Investigator
Masking Description: All clinical measurements were taken by a single blinded investigator (Periodontal Resident) while a single dental hygienist was responsible for prophylaxis and delivery of oral hygiene instructions to the study participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- water flosser (Experimental): patient will be provided with Waterpik Water Flosser and instructed to water floss around the implant once a day, preferably at nighttime
  Interventions: Device: comparing interdental floss to water flosser around dental implants
- dental floss (Active Comparator): patient will be instructed to floss with TePe Bridge and Implant Floss once a day, preferably at nighttime
  Interventions: Device: comparing interdental floss to water flosser around dental implants

INTERVENTIONS:
Device: comparing interdental floss to water flosser around dental implants — to determine the effectiveness in reducing the bleeding on probing (BOP) index around dental implants

SUMMARY:
The primary objective of this study was to compare two different interproximal devices, water flosser and dental floss around implants in several clinical parameters

DETAILED DESCRIPTION:
This study was a randomized, controlled clinical trial in a single center. All clinical measurements were taken by a single blinded investigator (Periodontal Resident) while a single dental hygienist was responsible for prophylaxis and delivery of oral hygiene instructions to the study participants. At each appointment 5 clinical parameters were recorded: Full Mouth Plaque Score (FMPS) and Quigley-Hein plaque index (QHI) of the implants after the use of a disclosing solution, Probing Depth (PD), Bleeding on Probing (BOP) of the study implants recorded at 6 sites (distobuccal, mid-buccal, mesiobuccal, distolingual, mid-lingual and mesiolingual) using a UNC 12 Colorvue probe and the width of the keratinized tissue (KT) at the buccal surface of the study implants. Randomization between the 2 groups was achieved using computerized randomization scheme (https://en.calc-site.com/randoms/grouping).

Group A (control): patients were instructed to floss with TePe Bridge and Implant Floss once a day, preferably at nighttime.

Group B (test): patients were provided with Waterpik Water Flosser and instructed to water floss around the implant once a day, preferably at nighttime.

During each appointment the study investigator measured clinical parameters and participants received oral hygiene instructions (OHI) and supportive periodontal therapy (SPT) by a single dental hygienist. Once the study was concluded patients were asked to fill-out a 2 question questionnaire inquiring how much they liked their interproximal device and how easy it was to be used in a scale 1 to 5.

ELIGIBILITY:
Inclusion Criteria:

* Patients that present with at least a single implant with a screw-retained crown
* Patients with general good health that do not have a condition contra-indicating routine dental treatment
* Patients that are compliant with the research protocol and methods
* Patients that have read, understood and signed the informed consent form

Exclusion Criteria:

* Patients with implants with cemented crowns
* Patients with any contact hypersensitivity to the related materials used in the study
* Tobacco users (vaping included)
* Patients unwilling to sign the informed consent form or follow the protocol of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-09-06 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Change in BOP (bleeding on probing) index around dental implants | All participants have been seen at baseline, follow-up 1 (interval ranging between 3 to 6 months)
  to determine the effectiveness of a waterfloss system compared to flossing in changing the bleeding on probing (BOP) index around dental implants. BOP is a sign of inflammation and is recorded as yes/no (yes for bleeding, no for absence of bleeding). BOP is a percentage calculated by dividing the number of bleeding sites divided by the total number of sites of each implant. A lower percentage indicates lower inflammation
Full Mouth Plaque Score (FMPS) | All participants have been seen at baseline, follow-up 1 (interval ranging between 3 to 6 months)
  to determine the differences between water flosser compared to flossing in changing the Full Mouth Plaque Score (FMPS). FMPS is a percentage calculated by dividing the number of plaque containing surfaces divided by the total number of available surfaces of each tooth/implant. A lower percentage indicates lower total plaque and means better plaque control
Quigley-Hein plaque index (QHI) around dental implants | All participants have been seen at baseline, follow-up 1 (interval ranging between 3 to 6 months)
  to determine the differences of a waterfloss system compared to flossing in (QHI) around dental implants. Quigley-Hein plaque index (QHI) is a scale 0 to 5.
  0 no plaque.
  1. separate flecks of plaque at the cervical margin of the tooth.
  2. a thin continuous band of plaque (up to one mm) at the cervical margin of the tooth.
  3. a band of plaque wider than one mm but covering less than one-third of the crown of the tooth.
  4. plaque covering at least one-third but less than two-thirds of the crown of the tooth.
  5. plaque covering two-thirds or more of the crown of the tooth.
  A lower number indicates better plaque control.
keratinized tissue (KT) around dental implants | All participants have been seen at baseline, follow-up 1 (interval ranging between 3 to 6 months)
  to evaluate the differences of a waterfloss system compared to flossing in the width of keratinized tissue (KT) around dental implants. KT is the stratified, squamous epithelium, that lines the vestibular and oral surfaces of the gingiva.
Probing Depth (PD) around dental implants | All participants have been seen at baseline, follow-up 1 (interval ranging between 3 to 6 months)
  to evaluate the differences of a waterfloss system compared to flossing in Probing Depth (PD) around dental implants. PD is the measurement of the depth of a sulcus by measuring in millimeters the distance from a gingival margin to the base of the sulcus with a calibrated periodontal probe.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Testori T, Del Fabbro M, Feldman S, Vincenzi G, Sullivan D, Rossi R Jr, Anitua E, Bianchi F, Francetti L, Weinstein RL. A multicenter prospective evaluation of 2-months loaded Osseotite implants placed in the posterior jaws: 3-year follow-up results. Clin Oral Implants Res. 2002 Apr;13(2):154-61. doi: 10.1034/j.1600-0501.2002.130205.x. PMID 11952735
- [Background] van Velzen FJ, Lang NP, Schulten EA, Ten Bruggenkate CM. Dental floss as a possible risk for the development of peri-implant disease: an observational study of 10 cases. Clin Oral Implants Res. 2016 May;27(5):618-21. doi: 10.1111/clr.12650. Epub 2015 Aug 11. PMID 26261052
- [Background] Montevecchi M, De Blasi V, Checchi L. Is Implant Flossing a Risk-Free Procedure? A Case Report with a 6-year Follow-up. Int J Oral Maxillofac Implants. 2016 May-Jun;31(3):e79-83. doi: 10.11607/jomi.4263. PMID 27183086
- [Background] Worthington HV, MacDonald L, Poklepovic Pericic T, Sambunjak D, Johnson TM, Imai P, Clarkson JE. Home use of interdental cleaning devices, in addition to toothbrushing, for preventing and controlling periodontal diseases and dental caries. Cochrane Database Syst Rev. 2019 Apr 10;4(4):CD012018. doi: 10.1002/14651858.CD012018.pub2. PMID 30968949
- [Background] Kelekis-Cholakis A, Rothney J. Maintenance of Implant Patients: A Narrative Review. Implant Dent. 2019 Apr;28(2):161-172. doi: 10.1097/ID.0000000000000837. PMID 30601226
- [Background] Magnuson B, Harsono M, Stark PC, Lyle D, Kugel G, Perry R. Comparison of the effect of two interdental cleaning devices around implants on the reduction of bleeding: a 30-day randomized clinical trial. Compend Contin Educ Dent. 2013 Nov-Dec;34 Spec No 8:2-7. PMID 24568169